CLINICAL TRIAL: NCT05211310
Title: Turkish Validity and Reliability of High Activity Arthroplasty Score After Total Knee Arthroplasty
Brief Title: Validity and Reliability of High-Activity Arthroplasty Score
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Afyonkarahisar Health Sciences University (Other)
Responsible Party: Principal Investigator, Emel Taşvuran Horata, PhD; Assistant Professor, Afyonkarahisar Health Sciences University
Other Study IDs: 2022/2
Record Dates: First submitted 2022-01-23; First posted 2022-01-27 (Actual); Last update posted 2023-12-27 (Actual); Status verified 2023-12

CONDITIONS: Arthroplasty Complications
Keywords: Knee Arthroplasty, Total; Validation Study; Questionnaire

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: High-Activity Arthroplasty Score (HAAS) — The questionnaire developed by Talbot et al. in 2010 consists of 4 sub-dimensions. 0-18 points can be obtained from the survey. High scores are associated with higher functional ability.
Other: Western Ontario and McMaster Universities osteoarthritis score (WOMAC) — It is used to evaluate disability in patients with hip and knee osteoarthritis. Each sub-dimension is standardized within the range of 0-100 points, with high scores indicating poor health.
Other: The Knee injury and Osteoarthritis Outcome Score (KOOS) — It is calculated between 0 and 100 points. 0 points indicate severe knee problem, 100 points no knee problem
Other: The Forgotten Joint Score-12 (FJS-12) — It evaluates how much an individual can forget an artificial joint during activities of daily living. A total of 100 points can be obtained. A high score is associated with the ability to forget.
Other: EQ-5D-5L — It is a questionnaire evaluating the quality of life. The higher the total score, the higher the quality of life.
Other: Numerical pain scale (NPS) — It is the numerical expression of perceived pain intensity. It is rated from 0-10 points. 10 points indicate the highest pain intensity, 0 points the absence of pain.

SUMMARY:
Patient-reported Outcome Measures (PROMs) used in total knee arthroplasty focus more on quality of life and pain. For this reason, individuals who can perform activities of daily living normally can get full points. There is a need for PROMs used in the assessment of higher functional skills. This study aimed to translate The High-Activity Arthroplasty Score (HAAS) into Turkish and to conduct a validity and reliability study of the Turkish version.

DETAILED DESCRIPTION:
Studies show that TKA practice has increased in the young population in recent years. Patient-reported Outcome Measures (PROMs) used in total knee arthroplasty focus more on quality of life and pain. For this reason, individuals who can perform activities of daily living normally can get full points. There is a need for PROMs used in the assessment of higher functional skills. This study aimed to translate The High-Activity Arthroplasty Score into Turkish and to conduct a validity and reliability study of the Turkish version. The adaptation of the questionnaire to Turkish in the study will be made according to the COSMIN and Reliability and Agreement Studies Reporting Guide. The construct validity, concurrent validity, reliability, and floor and ceiling effects of the questionnaire will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* To have undergone primary total knee arthroplasty for osteoarthritis at least 6 months ago,
* To be between the ages of 18-65.

Exclusion Criteria:

* Having orthopedic, neurological, cardiovascular, or cognitive problems that may affect physical performance,
* Presence of previous lower extremity surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Individuals who have undergone primary total knee arthroplasty surgery at least 6 months ago in the Orthopedics and Traumatology Outpatient Clinic will be included. Participants will be contacted via telephone.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
High-Activity Arthroplasty Score (HAAS) | 10 minutes
  It consists of 4 sub-dimensions (walking, running, climbing stairs and activity level). 0 (min. score) -18 points (max. score) can be obtained from the survey. Higher score is associated with more functional ability

CONTACTS AND LOCATIONS:
Overall Officials: EMEL TAŞVURAN HORATA, PhD, Principal Investigator — AFSU
Locations (2):
- Turkey (Türkiye) (2):
  - Afyonkarahisar Health Science University, Afyonkarahisar
  - Emel Taşvuran Horata, Afyonkarahisar

IPD SHARING:
Plan to Share IPD: No